CLINICAL TRIAL: NCT04092491
Title: Study of the IgA Repertoire During IgA Deposition Nephropathy.
Acronym: ERINA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Other Study IDs: 87RI19_0001
Record Dates: First submitted 2019-08-08; First posted 2019-09-17 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2019-05

CONDITIONS: Glomerulonephritis, IGA
Keywords: IgA nephropathy
MeSH Terms: conditions — Glomerulonephritis, IGA | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 1 blood sample during a consultation carried out as part of a medical follow-up:
  * 2 PAXgene RNA tubes of 2 ml each
  * 1 dry tube for creatinine and IgA assay
  * 1 tube of NFs (5ml)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1 blood sample: 1 blood sample during a consultation carried out as part of a medical follow-up:
  * 2 PAXgene RNA tubes of 2 ml each
  * 1 dry tube for creatinine and IgA assay
  * 1 tube of NFs (5ml)
  Interventions: Other: blood sample

INTERVENTIONS:
Other: blood sample — 1 blood sample during a consultation carried out as part of a medical follow-up:
  * 2 PAXgene RNA tubes of 2 ml each
  * 1 dry tube for creatinine and IgA assay
  * 1 tube of NFs (5ml)

SUMMARY:
IgA plays a major role in mucosal and systemic immunity but retains mysterious and ambivalent aspects. They can thus, depending on the situation, prove to be capable of triggering either a protective inflammatory response or, on the contrary, anti-inflammatory and inducing tolerance. Similarly, and for reasons that remain very poorly understood, they can be involved in pathologies where the immune system is itself an aggressor of the body and responsible for immunopathological lesions.

The investigator formulates the hypothesis that an inappropriate response of the mucosal immune system to one or more antigens leads to a synthesis of IgA of bad affinity favoring a deposit at the level of the mesangium. It seems important to verify this point by analyzing the IgA repertory of patients with N-IgA and comparing it to that of a control population.

DETAILED DESCRIPTION:
IgA plays a major role in mucosal and systemic immunity but retains mysterious and ambivalent aspects. They can thus, depending on the situation, prove to be capable of triggering either a protective inflammatory response or, on the contrary, anti-inflammatory and inducing tolerance. Similarly, and for reasons that remain very poorly understood, they can be involved in pathologies where the immune system is itself an aggressor of the body and responsible for immunopathological lesions.

the investigator formulates the hypothesis that an inappropriate response of the mucosal immune system to one or more antigens leads to a synthesis of IgA of bad affinity favoring a deposit at the level of the mesangium. It seems important to verify this point by analyzing the IgA repertory of patients with N-IgA and comparing it to that of a control population.

ELIGIBILITY:
Inclusion Criteria:

* Control population:

  * person between the ages of 18 and 55 (persons matched to age and sex (75% male) (N-IgA is more common in humans) free from any pathology.

oAbsence of proteinuria and hematuria on urine sample (search by strip).

* Patients with N-IgA

  * 40 patients with N-IgA whose diagnosis was confirmed by renal biopsy. These may be previously known patients who have not received treatment with corticosteroids or immunosuppressants for 12 months or new patients. The incidence of N-IgA is 20 patients per Mh; the number of incident patients with N-IgA is 10-15 per year in the nephrology department. The recruitment of 40 patients over 1 year is feasible.
  * Participant's written consent

Exclusion Criteria:

* Secondary or associated N-IgA (infection, malignant disease, inflammatory bowel disease,
* Rheumatic autoimmune disease or other;
* treatment with corticosteroids or immunosuppressants for less than 12 months.
* person on dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients with IgA nephropathy whose diagnosis was confirmed by renal biopsy
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2019-11-15 (Actual); Primary Completion 2020-11 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
To examine the immunoglobulins A | 1 year
  development of a technique for analyzing the repertoire of immunoglobulins

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Néphrologie, Limoges, France

IPD SHARING:
Plan to Share IPD: No